CLINICAL TRIAL: NCT00375492
Title: Effect on Weight Loss of Exenatide Versus Placebo in Subjects With Type 2 Diabetes Participating in a Lifestyle Modification Program
Brief Title: Effect on Weight Loss of Exenatide Versus Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H8O-US-GWBM
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Results first posted 2009-09-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; overweight; obesity; weight loss; exenatide; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Overweight; Obesity; Weight Loss | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: exenatide
- Group B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 5mcg or 10mcg, twice a day
  Other Names: Byetta
  Arms: Group A
Drug: placebo — subcutaneous injection, volume equivalent to exenatide dose, twice a day
  Arms: Group B

SUMMARY:
This trial is designed to compare the effects of twice-daily exenatide and twice-daily placebo on weight loss. This trial will evaluate overweight and obese subjects with type 2 diabetes who have inadequate glycemic control with metformin, sulfonylurea, or metformin plus a sulfonylurea. Subjects will be treated with exenatide or placebo in addition to their current oral antidiabetes agent regimen and participate in a lifestyle modification program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 6 months
* Have been treated with a stable dose of the following for at least 6 weeks prior to screening: *immediate or extended release metformin, or *a sulfonylurea, or *a fixed-dose sulfonylurea/metformin combination therapy
* Have an HbA1c of 6.6% to 10.0%, inclusive
* Have a Body Mass Index (BMI) of 25 kg/m^2 to 39.9 kg/m^2, inclusive

Exclusion Criteria:

* Are treated with any of the following excluded medications: *exogenous insulin, thiazolidinedione, or alpha-glucosidase inhibitor for more than 1 week within 6 weeks of screening; *Symlin injection at any time; * Byetta injection within 3 months of screening or discontinuation of therapy at any time due to adverse reaction; *drugs that directly affect gastrointestinal motility; *use of a weight loss drug (including those available over the counter) within 3 months of screening; *chronic (lasting longer than 2 weeks) systemic corticosteroids (excluding topical, intranasal, and inhaled preparations) by oral, intravenous, or intramuscular route within 2 months of screening
* Have conditions contraindicating metformin and/or sulfonylurea use
* Have had a change in lipid-lowering agents within 6 weeks of screening
* Have received glucagon-like peptide-1 (GLP-1) analogs, or dipeptidyl peptidase-IV inhibitors (DPP-IV inhibitors) or have previously participated in this study
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Malone, MD, Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - Research Site, Peoria, Arizona
  - Research Site, Jacksonville, Florida
  - Research Site, Orlando, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Spartanburg, South Carolina
  - Research Site, San Antonio, Texas
  - Research Site, Renton, Washington

REFERENCES:
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One randomized patient per group discontinued before receiving study drug. These patients are not included in the "started" category below.
Groups:
- Group A (Exenatide): exenatide 5mcg twice daily for 4 weeks, followed by exenatide 10mcg twice daily for 20 weeks
- Group B (Placebo): placebo (volume equivalent to exenatide injection) twice daily for 24 weeks
Period: Overall Study
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Started | 96 | 98
Completed | 70 | 72
Not Completed | 26 | 26
Not completed — Adverse Event | 4 | 5
Not completed — Entry Criteria Not Met | 0 | 1
Not completed — Loss of Glucose Control | 0 | 1
Not completed — Lost to Follow-up | 10 | 5
Not completed — Physician Decision | 0 | 4
Not completed — Protocol Violation | 6 | 3
Not completed — Sponsor Decision | 0 | 1
Not completed — Withdrawal by Subject | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Exenatide) | Group B (Placebo) | Total
Number analyzed (Participants) | 96 | 98 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 82 | 160
  >=65 years | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.52 (10.02) | 55.08 (8.97) | 54.81 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 61 | 121
  Male | 36 | 37 | 73
Baseline Body Weight [Mean (Standard Deviation); unit: kg] | 94.90 (16.52) | 96.16 (16.53) | 95.53 (16.05)
Baseline Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 4.67 (1.03) | 4.68 (0.90) | 4.68 (0.96)
Baseline Glycosylated Hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percent hemoglobin] | 7.74 (0.87) | 7.51 (0.82) | 7.62 (0.85)
Baseline High Density Lipoprotein (HDL) Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 1.18 (0.32) | 1.21 (0.31) | 1.20 (0.31)
Baseline Homeostatic Model Assessment-Beta Cell (HOMA-B) [Mean (Standard Deviation); unit: Percent beta-cell function] | 75.15 (81.20) | 70.72 (53.16) | 72.81 (67.65)
Baseline Homeostatic Model Assessment-Insulin Sensitivity (HOMA-S) [Mean (Standard Deviation); unit: Percent insulin sensitivity] | 49.72 (32.12) | 62.90 (41.07) | 56.68 (37.57)
Baseline Low Density Lipoprotein (LDL) Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 2.74 (0.88) | 2.78 (0.82) | 2.76 (0.85)
Baseline Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.15 (0.94) | 2.13 (1.00) | 2.14 (0.97)
Baseline Waist Circumference [Mean (Standard Deviation); unit: cm] | 109.64 (11.12) | 108.85 (12.10) | 109.24 (11.60)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Body Weight
Description: Change in body weight from baseline (Week 0) after 24 weeks of treatment (i.e., weight at week 24 minus weight at week 0). Body weight measured in kilograms (k).
Time Frame: Baseline, Week 24
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 70 | 72
kg | -6.16 (0.54) | -3.97 (0.52)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.0030, Mixed Model Repeated Measures

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Change in HbA1c from baseline (Week 0) after 24 weeks of treatment (i.e., HbA1c at week 24 minus HbA1c at week 0). HbA1c is measured as percent (%) of hemoglobin.
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: percent hemoglobin
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 70 | 71
percent hemoglobin | -1.21 (0.09) | -0.73 (0.09)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p < 0.0001, Mixed Model Repeated Measures

3. Secondary Outcome: Change From Baseline in 6-point Self Monitored Blood Glucose (SMBG) Profile at Week 24
Description: Change in SMBG at each of 6 time points throughout a day (blood glucose measurements before and 2 hours after the start of the morning, mid-day, and evening meals); week 24 compared to week 0 (i.e., SMBG at week 24 minus SMBG at week 0). Fasting Glucose measured in millimoles per liter (mmol/L).
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 69 | 72
mmol/L
  Morning Pre-Meal | -1.87 (0.17) | -1.20 (0.17)
  2 Hours Post Morning Meal | -2.67 (0.22) | -1.92 (0.22)
  Midday Pre-Meal | -1.40 (0.19) | -1.37 (0.19)
  2 Hours Post Midday Meal | -2.12 (0.21) | -1.51 (0.20)
  Evening Pre-Meal | -1.57 (0.19) | -1.32 (0.19)
  2 Hours Post Evening Meal | -3.09 (0.22) | -2.28 (0.23)

4. Secondary Outcome: Change From Baseline in Waist Circumference at Week 24
Description: Change in waist circumference from baseline after 24 weeks of treatment (i.e., waist circumference at week 24 minus waist circumference at week 0). Waist measured in centimeters (cm).
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 69 | 69
cm | -5.33 (0.71) | -4.18 (0.73)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.1985, Mixed Model Repeated Measures

5. Secondary Outcome: Ratio of Homeostatic Model Assessment-Beta Cell (HOMA-B) at Week 24 to HOMA-B at Baseline
Description: Ratio of HOMA-B at Week 24 to HOMA-B at baseline (Week 0). HOMA-B is a computer solved model used to predict the homeostatic concentrations which arise from varying degrees beta-cell deficiency. HOMA-B allows a quantitative assessment of the contributions of deficient beta cell function to the fasting hyperglycemia. HOMA-B is measured as a percent of the normal population (normal beta cell function = 100%, which is used as a reference in the calculation). The higher the percent the better for the participant.
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 68 | 76
Ratio | 1.46 (0.12) | 1.29 (0.10)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.1827, ANCOVA

6. Secondary Outcome: Ratio of Homeostatic Model Assessment-Insulin Sensitivity (HOMA-S) at Week 24 to HOMA-S at Baseline
Description: Ratio of HOMA-S at Week 24 to HOMA-S at baseline, week 0. HOMA-S is a computer solved model used to predict the homeostatic concentrations which arise from varying degrees of insulin sensitivity. HOMA-S allows a quantitative assessment of the contributions of insulin sensitivity to the fasting hyperglycemia. HOMA-S is measured as a percent of the normal population (normal insulin sensitivity = 100%, which is used as a reference in the calculation). The higher the percent the better for the participant.
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 68 | 76
Ratio | 1.08 (0.07) | 0.97 (0.06)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.1584, ANCOVA

7. Secondary Outcome: Change From Baseline in High Density Lipoprotein (HDL) Cholesterol at Week 24
Description: Change in HDL cholesterol from baseline after 24 weeks of treatment (i.e., HDL cholesterol at week 24 minus HDL cholesterol at week 0). HDL measured as mmol/L.
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 81 | 89
mmol/L | 0.02 (0.02) | 0.02 (0.02)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.8279, ANCOVA

8. Secondary Outcome: Change From Baseline in Low Density Lipoprotein (LDL) Cholesterol at Week 24
Description: Change in LDL cholesterol from baseline (Week 0) after 24 weeks of treatment (ie., LDL cholesterol at week 24 minus LDL cholesterol at week 0). LDL cholesterol measured in mmol/L
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 81 | 89
mmol/L | -0.06 (0.08) | -0.04 (0.07)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.8334, ANCOVA

9. Secondary Outcome: Change From Baseline in Total Cholesterol at Week 24
Description: Change in total cholesterol from baseline after 24 weeks of treatment (i.e., total cholesterol at week 24 minus total cholesterol at week 0). Total cholesterol measured in mmol/L.
Time Frame: baseline, week 24
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 81 | 89
mmol/L | -0.16 (0.10) | -0.03 (0.10)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.2881, ANCOVA

10. Secondary Outcome: Ratio of Triglycerides at Week 24 to Triglycerides at Baseline
Description: Ratio of triglyceride levels at Week 24 to triglyceride levels at baseline, Week 0 (ie., triglycerides at Week 24 divided by triglycerides at baseline, Week 0). Triglycerides measured in mmol/L.
Time Frame: baseline, Week 24
Population: Intent to Treat population
Measure: Geometric Mean (Standard Error); unit: Ratio
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 81 | 89
Ratio | 0.83 (0.04) | 0.92 (0.04)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.0654, ANCOVA

11. Secondary Outcome: Number of Participants With Hypoglycemic Events During the Study
Description: Number of participants experiencing one or more events of hypoglycemia at any point in the study
Time Frame: Baseline to 24 weeks
Population: Intent to Treat population
Measure: Number; unit: participants
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 96 | 98
participants | 33 | 30
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.728, Cochran-Mantel-Haenszel

12. Secondary Outcome: Rate of Hypoglycemic Events
Description: Overall rate of hypoglycemia, adjusted for 1 year (ie., events of hypoglycemia per participant per year).
Time Frame: 24 weeks
Population: Intent to Treat population
Measure: Least Squares Mean (Standard Error); unit: events per patient per year
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Number analyzed (Participants) | 96 | 98
events per patient per year | 7.14 (1.45) | 4.58 (1.43)
Statistical Analysis 1: Comparison: Group A (Exenatide) vs Group B (Placebo); Test type: Superiority or Other; p = 0.127, ANOVA

ADVERSE EVENTS:
Arm/Group | Group A (Exenatide) | Group B (Placebo)
Serious Adverse Events (participants affected / at risk) | 2 | 2
Other Adverse Events (participants affected / at risk) | 87 | 82
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Group A (Exenatide) | Group B (Placebo)
Gastroenteritis bacterial (Gastrointestinal disorders) | 1/96 | 0/98
Hypersensitivity (Immune system disorders) | 0/96 | 1/98
Nephrolithiasis (Renal and urinary disorders) | 1/96 | 0/98
Upper respiratory tract infection (Infections and infestations) | 0/96 | 1/98
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Group A (Exenatide) | Group B (Placebo)
Nausea (Gastrointestinal disorders) | 43/96 | 19/98
Diarrhea (Gastrointestinal disorders) | 18/96 | 21/98
Upper respiratory tract infection (Infections and infestations) | 17/96 | 17/98
Vomiting (Gastrointestinal disorders) | 21/96 | 9/98
Headache (Nervous system disorders) | 11/96 | 9/98
Constipation (Gastrointestinal disorders) | 9/96 | 10/98
Injection site bruising (General disorders) | 5/96 | 14/98
Nasopharyngitis (Infections and infestations) | 11/96 | 6/98
Back pain (Musculoskeletal and connective tissue disorders) | 4/96 | 8/98
Decreased appetite (Metabolism and nutrition disorders) | 6/96 | 6/98
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7/96 | 5/98
Cough (Respiratory, thoracic and mediastinal disorders) | 5/96 | 6/98
Contusion (Injury, poisoning and procedural complications) | 6/96 | 4/98
Dizziness (Nervous system disorders) | 5/96 | 5/98
Urinary tract infection (Infections and infestations) | 3/96 | 7/98
Myalgia (Musculoskeletal and connective tissue disorders) | 5/96 | 2/98
Dysgeusia (Gastrointestinal disorders) | 5/96 | 1/98
Injection site pruritus (General disorders) | 6/96 | 0/98
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1/96 | 5/98
Injection site erythema (General disorders) | 5/96 | 0/98
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5/96 | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.